CLINICAL TRIAL: NCT00894348
Title: EXEMPT: Prospective Factors Predicting Positive Yields on Biliary Brush Cytology During Endoscopic Retrograde Cholangio-pancreatography (ERCP)
Brief Title: Factors Predicting Positive Yields on Biliary Brush Cytology During Endoscopic Retrograde Cholangiopancreatography
Acronym: ERCP
Status: Completed | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Mansour Parsi, MD, MD, The Cleveland Clinic
Other Study IDs: IRB 09-032
Record Dates: First submitted 2009-05-05; First posted 2009-05-07 (Estimated); Last update posted 2017-03-30 (Actual); Status verified 2017-03

CONDITIONS: Biliary Stricture
Keywords: ERCP; Positive Biliary Brush Cytology

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
To determine factors associated with a positive yield of malignancy on biliary brush cytology obtained by ERCP.

DETAILED DESCRIPTION:
There are only 3 studies available that have tried to evaluate factors influencing the yield of brush cytology. Two of the 3 studied one parameter. The third study, which is also the largest, reported on 199 samples which the authors evaluated in a retrospect fashion. We plan to conduct a larger study assessing several other factors that have not been studied before. The study findings would help develop strategies to improve sensitivity of brush cytology specimens. This would ultimately result in more effective use of health care resources and improve patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* ERCP Patients

Exclusion Criteria:

* Non ERCP Patients

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing an ERCP for evaluation of biliary strictures
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2009-01; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
To determine factors associated with a positive yield of malignancy on biliary brush cytology obtained by ERCP determine the factors associated with a positive yield of malignancy on biliary brush cytology obtained by ERCP | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Mansour Parsi, M.D., Principal Investigator — Staff Physician
Locations (1):
- Cleveland Clinic Foundation, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No